CLINICAL TRIAL: NCT00679926
Title: A Phase IV Open Label Investigation of the Efficacy and Durability of Once Daily Antiretroviral Therapy With Kaletra and Viread in Antiretroviral Naïve Patients.
Brief Title: Kaletra and Viread in Antiretroviral Naïve Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Oklahoma State University Center for Health Sciences (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Johnny Stephens, Associate Professor, Oklahoma State University Center for Health Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Baker - 001
Record Dates: First submitted 2008-05-15; First posted 2008-05-19 (Estimated); Results first posted 2020-12-04 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: HIV Infections
Keywords: HIV; AIDS; HIV/AIDS; Treatment Naive
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — lopinavir-ritonavir drug combination; Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Once daily (Experimental): Patients taking 4 (four) lopinavir/ritonavir (200mg/50mg tablets) and 1 (one) tenofovir (300mg tablet) every 24 (twenty four) hours.
  Interventions: Drug: Once daily

INTERVENTIONS:
Drug: Once daily — Four tablets of lopinavir/ritonavir and one tablet of tenofovir given once daily
  Other Names: Kaletra; Viread

SUMMARY:
Once daily antiretroviral therapy with Viread (tenofovir DF, 300mg) plus Kaletra (LPV/r, 800mg/200mg) will be effective in suppressing and maintaining suppression of HIV RNA to <50 copies/ml in antiretroviral naïve patients through 48 weeks of therapy.

DETAILED DESCRIPTION:
This study is a phase IV prospective, open-label, controlled treatment protocol consisting of once daily Kaletra dosed at 800mg lopinavir with 200mg ritonavir in four combination tablets plus Viread dosed as 300 mg tenofovir DF. This will be a single site, multi-investigator, study for 48 weeks. Consecutive eligible patients will be enrolled into the study to reach the enrollment goal of 30 patients. Eligible patients will be identified and screened during routine initial or follow-up visits at the Internal Medicine Specialty Services Clinic. This clinic serves as the HIV/AIDS specialty care clinic and is a subdivision of the Department of Internal Medicine, Oklahoma State University Center for Health Sciences College of Osteopathic Medicine. The study site currently serves >700 persons living with HIV in northeast Oklahoma with four to five antiretroviral naïve patients seen each week.

Patients meeting all inclusion criteria will receive routine standard of care for our program as prescribed by the DHHS guidelines. Patients will have a Complete Blood Count (CBC), Complete Metabolic Profile (CMP), fasting lipid profile, CD4 count, HIV-1 RNA level, and other prescribed or indicated laboratory preformed at baseline and throughout the study as described in the Visits and Evaluations section of this protocol. All of the aforementioned laboratory tests will be performed at the Diagnostic Laboratories of Oklahoma, a division of Quest Diagnostics. Any antiretroviral resistance testing will be performed at Virologic Labs, Inc. Adherence will be assessed at discontinuation of the study and when indicated for evaluation of virologic failure by Memory Electronic Monitoring Systems caps and pharmacy refill data. Patients will be monitored at each study visit for tolerability and adverse events. Patients who develop a study related Grade 1 or 2 Adverse Events (Aes) may continue the study. Those who develop Grade 3 or 4 AEs will have study medications discontinued. Patients with asymptomatic elevations of triglyceride or Low Density Lipoprotein (LDL) cholesterol levels may be treated with appropriate lipid lowering therapy at the investigators discretion.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients >18 years of age with documented HIV-1 infection
2. Naïve to antiretroviral therapy
3. Able and willing to provide written informed consent
4. No CD4 restriction
5. HIV-1 RNA levels >5000 c/mL
6. Female patients must meet these additional criteria

   1. Non-childbearing potential
   2. Negative serum pregnancy test at screen
   3. Willingness to abstain from sexual intercourse or use double barrier contraception

Exclusion Criteria:

1. Presence of any of the following:

   1. Aminotransferases >3xULN
   2. Hemoglobin concentration <8.0g/dl
   3. Absolute neutrophil count <800 cells/cubic mm
   4. Platelet count <50,000 cells/cubic mm
   5. Acute illness, or an acute illness ≤7 days
   6. Presence of Opportunistic Infection, or an OI within 30 days of screening
   7. Acute or chronic active Hepatitis B
   8. Hepatitis C
   9. Creatinine Clearance <50 mL/min
2. Pregnant or breast-feeding women
3. Presence of any illness, physical or behavioral conditions (i.e., substance abuse, excluding cannabis) that will impair the patient's ability participate
4. Patient who, in the opinion of the investigator, will be unlikely to complete the study protocol and adhere to the study drug regimens
5. Concurrent use of medications that may potentially interact with study medications including: astemizole, terfenadine, rifampin, dihydroergotamine, ergonovine, ergotamine, methylergonovine, cisapride, St. John's wort, lovastatin, simvastatin, pimozide, midazolam, triazolam, adefovir, cidofovir, acyclovir, ganciclovir, and valganciclovir.
6. Patient suffers from a serious medical condition that may in the opinion of the investigator compromise his or her safety.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-05; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Damon Baker, D.O., Principal Investigator — Oklahoma State University Center for Health Sciences
Locations (1):
- OSU Internal Medicine Specialty Clinic, Tulsa, Oklahoma, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was July 2009 to January 2011 and was completed at the Internal Medicine Specialty Clinic at OSU-CHS.
Pre-assignment Details: There are no significant events prior to enrollment. Patients had to be naive to HIV therapy prior to treatment drug.
Groups:
- Single Treatment Arm: Patients taking lopinavir/ritonavir and tenofovir once daily.
  Lopinavir/ritonavir and tenofovir : Four tablets of lopinavir/ritonavir and one tablet of tenofovir given once daily
Period: Overall Study
Arm/Group | Single Treatment Arm
Started | 15
Completed | 2
Not Completed | 13

BASELINE CHARACTERISTICS:
Arm/Group | Single Treatment Arm
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: To Assess the Efficacy of Once Daily Antiretroviral Therapy With Viread 300mg and Kaletra 800mg/200mg in Suppressing HIV RNA Levels to <50 Copies/ml in Antiretroviral naïve Patients.
Description: To assess the efficacy of once daily antiretroviral therapy with Viread 300mg and Kaletra 800mg/200mg in suppressing HIV RNA levels to <50 copies/ml in antiretroviral naïve patients. This will be done by the proportion of patients with plasma HIV-1 RNA levels M 50 copies/ml at the end of 48 weeks of therapy.
Time Frame: 4, 8, 12, 16, 24, 32, 40, and 48 weeks
Population: The study was terminated due to lack of enrollment and data were not collected from 13 out of 15 participants.
Arm/Group | Single Treatment Arm
Number analyzed (Participants) | 0

2. Secondary Outcome: Proportion of Patients With <400copies/ml
Description: Proportion of patients with <400copies/ml will be done by determining plasma HIV-1 RNA levels
Time Frame: 4,8, and 12 weeks
Population: The study was terminated due to lack of enrollment and data were not collected from 13 out of 15 participants.
Arm/Group | Once Daily
Number analyzed (Participants) | 0

3. Secondary Outcome: Review Virologic Response to Assess Rate of Viral Decline.
Description: Review virologic response to assess rate of viral decline through CD4 count at baseline and throughout the study.
Time Frame: weeks 4, 8, 12, 16, and 24
Population: The study was terminated due to lack of enrollment and data were not collected from 13 out of 15 participants.
Arm/Group | Single Treatment Arm
Number analyzed (Participants) | 0

4. Secondary Outcome: Proportion of Patients With <50 Copies/ml HIV-1 RNA
Description: Proportion of patients with <50 copies/ml HIV-1 RNA through evaluation of patients Plasma HIV-1 RNA levels
Time Frame: at weeks 4, 8, 12, 16, 24, 32, 40, and 48
Population: The study was terminated due to lack of enrollment and data were not collected from 13 out of 15 participants.
Arm/Group | Single Treatment Arm
Number analyzed (Participants) | 0

5. Secondary Outcome: Change From Baseline CD4 Counts
Description: CD4 count done at baseline and throughout the study.
Time Frame: at weeks 4, 8, 12, 16, 24, 32, 40, and 48
Population: The study was terminated due to lack of enrollment and data were not collected from 13 out of 15 participants.
Arm/Group | Single Treatment Arm
Number analyzed (Participants) | 0

6. Secondary Outcome: Time to Virologic Failure.
Description: Virologic failure is defined by any of the following: 1) <1 log10 decline in HIV RNA by week 8 of therapy; 2) failure to achieve <50 c/mL by week 24; 3) HIV RNA> 500 c/ML on two consecutive occasions (less than 30 days apart), with no evidence of suppression after adherence counseling. When HIV RNA levels are obtained >500 copies/mL it will be repeated within 2 weeks. If after adherence counseling, HIV RNA demonstrates > 1 log 10 decline but remains >500, the patient will receive a final adherence counseling session and have his/her HIV RNA measure repeated at day 30: if a third consecutive HIV RNA remains 500 c/mL the patient will be removed from study, if <500c/mL the patient will remain on study
Time Frame: Week 48
Population: The study was terminated due to lack of enrollment and data were not collected from 13 out of 15 participants.
Arm/Group | Single Treatment Arm
Number analyzed (Participants) | 0

7. Secondary Outcome: Tolerability and Adverse Events.
Description: Adverse events and safety parameters are monitored for ll subjects for the duration of the study. Toxicities and adverse events will be graded using the modified ACTG toxicity ratings scale. Study drugs may be interrupted for safety reasons and/or based on grade of toxicity/adverse event.
Time Frame: 48 weeks
Population: The study was terminated due to lack of enrollment and data were not collected from 13 out of 15 participants.
Arm/Group | Single Treatment Arm
Number analyzed (Participants) | 0

8. Secondary Outcome: Change From Baseline Fasting Total Cholesterol and Fasting Triglyceride Levels.
Description: Change from baseline fasting total cholesterol and fasting triglyceride levels will be measured by fasting lipid panels taken at baseline and at various timepoints.
Time Frame: 48 weeks
Population: The study was terminated due to lack of enrollment and data were not collected from 13 out of 15 participants.
Arm/Group | Once Daily
Number analyzed (Participants) | 0

9. Secondary Outcome: Characterize Adherence Rates for This Therapeutic Regimen by the Use of Medication Electronic Monitoring Systems (MEMS) Caps.
Description: The medication event monitoring system (MEMS) is a cap that fits on standard medicine bottles and records the time and date each time the bottle is opened and closed.
Time Frame: 48 weeks
Population: The study was terminated due to lack of enrollment and data were not collected from 13 out of 15 participants.
Arm/Group | Single Treatment Arm
Number analyzed (Participants) | 0

10. Secondary Outcome: Characterize Adherence Rates for This Therapeutic Regimen by Use of Pharmacy Refill Records.
Description: Characterize adherence rates for this therapeutic regimen by use of pharmacy refill records is assessed by an examination of pharmacy refill data for patients.
Time Frame: 48 weeks
Population: The study was terminated due to lack of enrollment and data were not collected from 13 out of 15 participants.
Arm/Group | Once Daily
Number analyzed (Participants) | 0

11. Secondary Outcome: Assess Genotypic Changes in Patients With Virologic Failure.
Description: At time of virologic failure genotypes will be performed on baseline and failure isolates; phenotypic testing will be performed on failure isolates to examine LPV susceptibility.
Time Frame: 48 weeks
Population: The study was terminated due to lack of enrollment and data were not collected from 13 out of 15 participants.
Arm/Group | Once Daily
Number analyzed (Participants) | 0

12. Secondary Outcome: Assess Lopinavir Trough Levels in Patients Failing to Obtain Virologic Suppression.
Description: Assess lopinavir trough levels in patients failing to obtain virologic suppression by measuring lopinavir trough level
Time Frame: 48 weeks
Population: The study was terminated due to lack of enrollment and data were not collected from 13 out of 15 participants.
Arm/Group | Once Daily
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Single Treatment Arm
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No